CLINICAL TRIAL: NCT01458457
Title: Life Quality and Mental State in Patients With Breast Cancer - a Randomized Study
Brief Title: Life Quality and Mental State in Patients With Breast Cancer
Acronym: BBK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Azienda Sanitaria de Sudtirol, Hospital Meran, Meran, Italy (Unknown)
Responsible Party: Principal Investigator, Claudia M. Witt, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBK
Record Dates: First submitted 2011-10-21; First posted 2011-10-24 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator)
  Interventions: Other: Individualized usual care
- Usual Care + Complementary Medicine (Active Comparator)
  Interventions: Other: Individualized complementary medicine treatment; Other: Individualized usual care

INTERVENTIONS:
Other: Individualized complementary medicine treatment — An individual treatment plan will be made for each patient that includes one to all of the following treatments: acupuncture, traditional Chinese herbal medicine, enzyme therapy, nutrition advise, Healing Touch, homoeopathy, hyperthermia treatment, infusions, laser therapy, lymphatic drainage, manual therapy, mistel therapy, neural therapy, orthomolecular therapy, osteopathy, phytotherapy, shiatsu
  Arms: Usual Care + Complementary Medicine
Other: Individualized usual care — Patients get usual care from their general practitioners/specialized physicians

SUMMARY:
Randomized pragmatic trial to evaluate the comparative effectiveness regarding disease specific quality of life of an individualized additional complementary medicine treatment in addition to usual care with usual care only in 280 women with breast cancer

ELIGIBILITY:
Inclusion Criteria:

* diagnosed breast cancer
* current usual care treatment
* willing to refrain from complementary treatment for 6 months in case of randomization into the usual care group
* informed consent

Exclusion Criteria:

* complementary treatment at the Hospital Meran in the last 6 months
* no German or Italian language ability
* participation in other study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) | 6 months

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy-Breast quality of life instrument (FACT-B) | 3 months
Subscales of the Functional Assessment of Cancer Therapy - General (FACT-G): physical well-being, social/family well-being, emotional well-being, functional well-being) | 3, 6 months
Subscale for Breast Cancer of the Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) | 3, 6 months
Pain, quality of sleep, and nausea (single items of the FACT-B) | 3, 6 months
Functional Assessment of Chronic Illness Therapy-Fatigue | 3, 6 months
Survival without relapse | 6 months
Quality of Life (SF-12 Health Survey) | 3, 6 months
Undesirable Effects and Interactions | 6 months
Goal Attainment Scale | 3 months
  This outcome measures will only be assessed in the complementary medicine arm
Used complementary Therapies and their frequency | 6 months
  This will only be assessed in the complementary medicine arm
Expectations at Baseline | Baseline
  This will only be assessed in the complementary medicine group
Satisfaction and patient-reported effectiveness | 3, 6 months
  This will only be assessed in the complementary medicine arm
Survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M Witt, Prof. Dr. med., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Meran Hospital - Dienst fuer Komplementaermedizin, Meran, Italy

REFERENCES:
- [Result] Witt CM, Ausserer O, Baier S, Heidegger H, Icke K, Mayr O, Mitterer M, Roll S, Spizzo G, Scherer A, Thuile C, Wieser A, Schutzler L. Effectiveness of an additional individualized multi-component complementary medicine treatment on health-related quality of life in breast cancer patients: a pragmatic randomized trial. Breast Cancer Res Treat. 2015 Jan;149(2):449-60. doi: 10.1007/s10549-014-3249-3. Epub 2015 Jan 3. PMID 25555830